CLINICAL TRIAL: NCT01786304
Title: Effect of Sacral Nerve Stimulation on Enteric Nervous System
Acronym: ENS-3
Status: Completed | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Collaborators: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2012/091/HP
Record Dates: First submitted 2013-02-05; First posted 2013-02-07 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-12

CONDITIONS: Fecal Incontinence
Keywords: Fecal incontinence, sacral nerve stimulation
MeSH Terms: conditions — Fecal Incontinence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — colonic biopsies
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Fecal incontinence: Patient with fecal incontinence and referred for a treatment with sacral nerve stimulation
  Interventions: Procedure: Sacral nerve stimulation

INTERVENTIONS:
Procedure: Sacral nerve stimulation — implantation of a stimulation electrode in one of the S2-S3-S4 sacral hole then connected to a subcutaneous stimulator for permanent stimulation of the sacral nerve

SUMMARY:
Sacral nerve stimulation (SNS) is a new therapeutic option to treat fecal incontinence, although its mecanims of action remains poorly understood. The investigators hypothtized that SNS could act on enteric nervous system (ENS). To verify this hypothesis, the investigators will collect biopsy samples from patients implanted for SNS, and assess whether SNS induces changes in ENS.

DETAILED DESCRIPTION:
Sacral nerve stimulation (SNS) is a new therapeutic option to treat fecal incontinence. Its efficacy yields 80% approximately, but its mecanims of action remains poorly understood. In particular, SNS does not restore anal squeezing contraction nor it increase anal tone. Recently, using a porcine model, it was shown that SNS changed colonic permeability, suggesting that SNS may activate the enteric nervous system (ENS).

The investigators hypothtized therefore that SNS could act on enteric nervous system (ENS).

To verify this hypothesis, the investigators will collect biopsy samples from patients before and after implantation for SNS. The investigators will assess whether SNS induces changes in ENS, and if this is correlated to SNS efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Fecal incotinence
* refractory to medial treatment
* Eligible to a treatment with sacral nerve stimulation

Exclusion Criteria:

* age < 18 yo
* age < 75 yo
* anal defect > 120°
* bilateral interruption of the bulbo-cavernous reflex
* patient not able to speack and understand the French Language
* patient not affilated to the French healthcare system
* pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with fecal incontience refractory to standard medical treatment
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2013-01; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Number of neurons producing vasoactive intestinal peptide (VIP) | 6 months
  Number of neurons producing vasoactive intestinal peptide (VIP) by immunochemistry

SECONDARY OUTCOMES:
Number of cholinergic neurons | 6 months
  Number of cholinergic neurons by immunochemistry

OTHER OUTCOMES:
Fecal incontinence score | 6 months
  Measured using the Cleveland Clinic score
Quality of life | 6 months
  measured using the FIQL score that has been validated in french

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Gourcerol, MD, PhD, Principal Investigator — Rouen University Hospital, France
Locations (2):
- France (2):
  - Rouen University Hospital, Rouen, Normandy
  - Nantes University Hospital, Nantes, Pays de Loire